CLINICAL TRIAL: NCT00412815
Title: The Effects of Exercise Training on Insulin Resistance in Patients With Coronary Artery Disease and Insulin Resistance, the Exercise, Coronary Artery Disease and Insulin Resistance (EXCADIR) Randomized Controlled Trial
Brief Title: Exercise Training, Insulin Resistance and Coronary Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R-99-004
Record Dates: First submitted 2006-12-14; First posted 2006-12-18 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease; Glucose Intolerance
Keywords: insulin sensitivity; coronary artery disease; exercise training
MeSH Terms: conditions — Coronary Artery Disease; Glucose Intolerance; Insulin Resistance | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise training

SUMMARY:
The purpose of this study was to determine the effects of exercise training on insulin resistance in subjects with coronary artery disease independent of changes in weight, diet, or the effect of an acute bout of exercise. We hypothesized that subjects with CAD and high normal or impaired glucose tolerance performing 12 weeks of aerobic exercise training while on a non weight-reducing diet, would have a greater decrease in insulin resistance than controls measured at 72 hours following their last bout of exercise.

DETAILED DESCRIPTION:
Objectives To determine the effects of exercise training on insulin resistance in CAD subjects without diabetes, independent of changes in weight, diet, or the effect of acute exercise.

The study was approved by the Research Ethics Review Boards at London and Hamilton. All participants provided written and verbal informed consent.

Inclusion Criteria The study population will include men and women over 18 years of age identified from the practices of local cardiologists, whose fasting plasma glucose concentration is 5.4-7.7 mmol/L, and who had confirmed CAD (diagnosed on the basis of a previous myocardial perfusion study or cardiac catheterization, or a history of a myocardial infarction or coronary artery angioplasty or coronary artery bypass surgery).

Exclusion Criteria Individuals will be excluded if they had known type 1 or 2 diabetes, clinical heart failure, uncorrected significant valvular or congenital heart disease, significant obstructive pulmonary disease (forced expiratory volume in 1 sec / forced vital capacity < 0.5), uncontrolled hypertension (blood pressure > 220 / 120 mm Hg), participation in a regular exercise program within the preceding three months, inability to perform exercise training, atrial fibrillation, a permanent pacemaker or regularly used corticosteroid. Individuals who had experienced a myocardial infarction, unstable angina, coronary artery bypass graft surgery, or coronary artery angioplasty within the 3 months prior to study entry were also excluded. Furthermore, individuals were excluded if their run-in phase fasting blood glucose was < 5.4 mmol/L or > 11.1 mmol/L at 2 hours following the 75 gram oral glucose load.

Screening Visit Individuals who satisfied the above criteria underwent a screening visit comprising a full explanation of the study, appropriate history and physical evaluation by one of the study physicians (NGS or RSM). Height (m), weight (kg), waist and hip circumference (cm), and percentage body fat using bioelectrical impedance were measured. A 75g OGTT, using fasting and 2 hour samples, was then performed following an overnight (≥12 hour) fast. Participants satisfying the study selection criteria subsequently entered the run-in-phase.

Run-in Phase The study dietician assessed all participants and administered a 24-hour food recall and semi-quantitative food frequency questionnaire. An individualized isocaloric AHA Phase I diet with written and verbal instructions was prescribed to each patient. Participants were also taught how to complete a three-day measured food record. The purpose of the run-in phase was to have participants follow an AHA Phase I diet for at least 3 weeks, therefore the duration of the run-in phase was zero, three, or six weeks depending on the patient's current diet as determined by the study dietician. At the midpoint of the run-in phase, food records were reviewed to ensure completeness of food descriptions, preparation methods, portion sizes, and additional dietary counseling was provided as required. Baseline testing was carried out on completion of the run-in diet phase.

Baseline Testing Measurements included OGTT, waist circumference, body fat, a symptom-limited CET with measurement of oxygen consumption, and the 3-hour FSIGT to determine insulin resistance. The CET was performed on the first day of the subject's baseline assessments. On the morning of the CET participants were instructed to take their usual medications, to eat only a light breakfast and to abstain from caffeine. VO2 was continuously measured throughout the CET and the peak VO2 served as the index of exercise capacity. The CET was conducted according to accepted guidelines.

The FSIGT was performed 72 hours following the baseline CET after an overnight fast. Intravenous cannulas were placed in the antecubital vein of each arm. A glucose injection (500mg/kg as a 50% solution) was given over 1 minute starting at time 0 minutes. Blood samples for the determination of glucose and insulin were taken at -10, -5, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 19, 22, 24, 25, 27, 30, 40, 50, 60, 70, 80, 90, 100, 120, 140, 160, and 180 minutes following the conclusion of the glucose infusion. Twenty minutes following the start of the intravenous glucose, 0.04 U/kg of human insulin (Novolin R) was injected. Insulin sensitivity was determined using the validated MINMOD-IS technique. The MINMOD-IS determination was made by one of the investigators (DF) blinded to the patient's group allocation.

After satisfactory completion of baseline testing, participants were randomized to either 12-weeks of ET or UA. Randomization was computer generated following a non-blocked strategy and delivered using sealed envelopes. All individuals recording the outcome measurements were blinded to the group allocations of the participants. In order to maintain a stable weight throughout the study and in addition to the well-controlled AHA Phase I diet, ET participants underwent supervised weekly weigh-ins and were prescribed supplemental food in proportion to the AHA Phase I diet by the study dietician if weight loss of ≥ 1 kg occurred on two consecutive weekly supervised weigh-ins.

Participants in the UA group were instructed to continue their usual activity and to follow the AHA Phase I diet that was used in the week prior to randomization and to weigh themselves weekly on the same home scale, first thing in the morning with minimal attire. Participants contacted the study dietician if ≥ 1 kg weight change occurred over two weeks. Appropriate dietary adjustments were then made to ensure a stable weight. The ET group was prescribed exercise 4 times/week for 12 weeks. This exercise comprised walking, stationary cycling or treadmill exercise for 40 minutes per session at 75% of their baseline CET peak heart rate with 5-minute warm up and cool down periods. Participants were taught how to monitor their heart rate during exercise and to adjust their exercise intensity accordingly. Two of these sessions were conducted under supervision at the Hamilton Health Science Cardiac Rehabilitation Program while the remaining sessions were carried out at home.

Ten to 12 weeks following randomization all participants underwent endpoint assessments, which comprised the same testing as baseline. These assessments were OGTT & clinical evaluation (week 11), CET (week 12) and FSIGT (72 hours after CET). All participants were instructed not to perform any exercise training between the final CET and FSIGT.

Statistical Issues Fifty subjects overall were required to satisfy the study's sample size assumptions that at least a 15% decrease of insulin resistance with ET compared to UA could be demonstrated with 80% power, a 2-tailed alpha error of 5%, and a potential 20% loss to follow up rate. A Wilcoxon Rank-Sum Test was used to compare the change in MINMOD-IS over the course of the study between the ET and UA groups. Remaining analyses comparing outcomes between the ET and UA groups utilized independent t-tests for continuous data with normal distributions and Wilcoxon Rank-Sum Tests for continuous data that were not normally distributed. Regression analyses were done to evaluate relationships between the change of MINMOD-IS during the study and other important study variables such as changes in weight and peak VO2. Analyses were deemed significant if a two-tailed P-value of < 0.05 was achieved. All values are reported as the mean +/- standard deviation unless otherwise specified.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18 years of age
* fasting plasma glucose concentration 5.4-7.7 mmol/L
* confirmed CAD (diagnosed on the basis of a previous myocardial perfusion study or cardiac catheterization, or a history of a myocardial infarction or coronary artery angioplasty or coronary artery bypass surgery).

Exclusion Criteria:

* known type 1 or 2 diabetes
* clinical heart failure
* uncorrected significant valvular or congenital heart disease
* significant obstructive pulmonary disease (forced expiratory volume in 1 sec / forced vital capacity < 0.5)
* uncontrolled hypertension (blood pressure > 220 / 120 mm Hg)
* participation in a regular exercise program within the preceding three months
* inability to perform exercise training, atrial fibrillation
* a permanent pacemaker
* regularly used corticosteroid
* recent (< 3 months) myocardial infarction, unstable angina, coronary artery bypass graft surgery, or coronary artery angioplasty
* run-in phase fasting blood glucose was < 5.4 mmol/L or > 11.1 mmol/L at 2 hours following the 75 gram oral glucose load.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 1998-11-25 (Actual); Primary Completion 2000-06-09 (Actual); Study Completion 2000-06-09 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity

SECONDARY OUTCOMES:
Exercise capacity

CONTACTS AND LOCATIONS:
Overall Officials: Robert S McKelvie, MD, Principal Investigator — McMaster Univesrity
Locations (1):
- Hamilton Health Sciences Centre, Hamilton, Ontario, Canada